CLINICAL TRIAL: NCT02554838
Title: How to Act on the Mobility Restriction Linked to Senior's Phobia of Falling
Acronym: PACTE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K140702; 2015-A00400-49 (Other: ID RCB)
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Specific Phobia; Fear of Falling
Keywords: Specific phobia; Fear of Falling; Life-space area
MeSH Terms: conditions — Phobia, Specific | interventions — Exercise; Rehabilitation; Home Care Services; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation (Active Comparator): Rehabilitation :
  * Physical activity
  * Home assessment and modification
  Interventions: Other: Physical activity; Other: Home assessment and modification
- Rehabilitation and CBT (Experimental): Rehabilitation associated with cognitive behavioral therapy (CBT) :
  * Physical activity
  * Home assessment and modification
  * Cognitive behavioral therapy
  Interventions: Other: Physical activity; Other: Home assessment and modification; Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Other: Physical activity — Participants receive a weekly individual session of physical activity during 8 consecutive weeks conducted by a licensed physical therapist and focusing on muscle strengthening, flexibility, gait and balance retraining.
  Other Names: Rehabilitation
Other: Home assessment and modification — Two home-based sessions of modification of the home environment by a licensed rehabilitation therapist, in order to increase the aera of mobility, the frequency of moving in this aera and the independence to move.
  Other Names: Home Care Services
Behavioral: Cognitive behavioral therapy — Participants receive during 8 consecutive weeks a weekly individual sessions of CBT and a booster session one month later conducted by a psychologist specialized in CBT focusing on : functional analysis, education about treatment and anxiety, relaxation training and progressive exposure in imagination then in vivo.
  Other Names: Specific phobia; Fear of Falling; Life-space area
  Arms: Rehabilitation and CBT

SUMMARY:
This project aims to determine the respective impacts of two routine care regarding phobic of falling seniors on the mobility restriction. The investigators used a monocentric, randomized and controlled research according to two parallel groups : physical activity, home assessment and modification (rehabilitation group) versus physical activity, home assessment and modification with cognitive behavioral therapy (CBT) (rehabilitation and CBT group). The investigators will assess the efficacy of usual care (rehabilitation group) and the supplementary benefit of CBT (rehabilitation and CBT group) with the Life Space Assessment.

DETAILED DESCRIPTION:
The fear of falling affects about 20% of seniors living at home, having fallen beforehand or not. Its repercussions, like the premature decline of physical capacities, the decrease in quality of life, the loss of independence and the independent risk of falling are well known. They appear mediated by a restriction of mobility when the phobias of falling take place. Indeed, when a phobia of falling occurs, the person limits her moving to avoid the situations confronting her to the object of her fear - in this case, the fall. However, individuals going outdoors less frequently or moving through smaller life-space areas likely have poorer health and function, and coexisting lower levels of physical activity. Thus increasing life-space area may provide important health benefits in elderly people phobic of the fall.

The usual cares of the phobia of falling are physical activity, home assessment and modification with or without CBT programs. Their efficacy on the increase in mobility has not been properly assessed. One of the priorities is to assess these programs with some tools reporting improvement in mobility and independence.

The Life-Space Assessment (LSA) questionnaire of the Alabama and Birmingham Study of Aging can measure the evolution of the life-space area in an appropriate way, i.e. the spatial area in which a person commonly acts. This 20-item assessment captures the life-space mobility of individuals in five successive areas or life-space (LS) levels (from within the home to outside of town). Subjects are asked the frequency with which they moved in each of the five areas over the past four weeks, and if any assistance (from other persons or with equipment) or no assistance was required. A composite life space score (LSC, range: 0-120) is calculated combining information on the life space level, the degree of independence, and the frequency. Higher scores indicate greater life space. The reliability and construct/criterion validity of this questionnaire translated into French has been published.

The purpose of this study is to compare the effectiveness on an aera of mobility, measured using LSC on three months program combinating physical activity, home assessment and modification (rehabilitation group), versus a program combinating physical activity, home assessment and modification, and CBT (rehabilitation and CBT group) of the senior older than 70, suffering from phobia of falling and living at home.

After the initial study assessment, each participant will benefit during 8 consecutive weeks of a weekly individual session of physical activity, 2 home-based sessions of modification of the home environment and, moreover, for the patients of the rehabilitation and CBT group, a weekly session of individual CBT during the 8 consecutive weeks of the program and a booster session one month later.

Participation in this study will last up to 8 months. LSC will be tested in both groups before, immediately after, 3 and 6 months after completion of the intervention period to explore the benefit of each intervention.

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* to have a phobia of the fall (according to diagnostic criteria Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) of specific phobia)

Exclusion Criteria:

* Living in a nursing home
* Depression (Mini-Geriatric Depression scale score equal 1 or above)
* Cognitive impairment
* Medical conditions that would be incompatible or limit compliance with the study requirements
* Unable to walk even with assistance
* Patient in a period of exclusion relative to a biomedical study
* Patient's refusal of participation

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Life-space mobility assessed by the LSC (a composite score of the Life-Space Assessment which reflects the distance, frequency and level of independence of movement during the 4 weeks preceding the assessment) at 5 months. | Baseline, 5 months (3 month follow-up)
  For each life-space level (bedroom (score 0), other rooms (1), outside home (2), neighborhood (3), town (4), beyond town (5)), participants were asked how many days a week they attained that level (frequency; <1×/week (score 1), 1-3x/week (2), 4-6x/week (3), daily (4)) and whether they needed help from another person or from assistive devices (assistance; no assistance (score 2), equipment only (1½), personal assistance needed (1)). The LSC ranging from 0 to 120 was calculated based on life-space level *degree of independence in achieving each level * frequency of attaining each level, and then summed for all levels, with higher score representing greater mobility.

SECONDARY OUTCOMES:
Change from baseline in Life-space frequency (a composite score of the Life-Space Assessment which reflects the distance and frequency of movement during the 4 weeks preceding the assessment) at 2, 5 and 8 months. | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  The life-space frequency ranging from 0 to 60 was calculated based on life-space level score * frequency score at respective level, and then summed, with higher score representing greater mobility.
Change from baseline in Assisted life-space (a score of the Life-Space Assessment which indicating the highest level of life-space attained using the help of assistive devices if needed but not the help of another person) at 2, 5 and 8 months. | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  The assisted life-space ranging from 0 to 5 was calculated based on life-space level score attained using the help of assistive devices if needed but not the help of another person.
Change from baseline in Life-space mobility assessed by the LSC (a composite score of the Life-Space Assessment which reflects the distance, frequency and level of independence of movement during the 4 weeks preceding the assessment) at 2, 5, 8 months. | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  For each life-space level (bedroom (score 0), other rooms (1), outside home (2), neighborhood (3), town (4), beyond town (5)), participants were asked how many days a week they attained that level (frequency; <1×/week (score 1), 1-3x/week (2), 4-6x/week (3), daily (4)) and whether they needed help from another person or from assistive devices (assistance; no assistance (score 2), equipment only (1½), personal assistance needed (1)). The LSC ranging from 0 to 120 was calculated based on life-space level *degree of independence in achieving each level * frequency of attaining each level, and then summed for all levels, with higher score representing greater mobility.
Number of falls and injurious falls | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  Falls were defined as "unintentionally coming to rest on the ground, floor, or other lower level" and collected by face-to-face interview of subjects.
  Fall events were classified as resulting in "serious" injury if the fall resulted in a fracture, head injuries requiring hospitalisation, joint dislocation, serious sprain, other serious joint injuries, admission to hospital or if any wounds needed stitches (sutures), "moderate" injury if bruising, not serious sprains, cuts, abrasions, or reduction in physical function for at least three days resulted or if the participant sought medical help, and "no" injury.
Fear of falling | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  Fear of Falling will be measured using the Falls Efficacy Scale-International (FES-I) , a self-report questionnaire of 16 items measuring level of concern about falling during 16 activities of daily living. Minimum score 16, maximum score 64.
Use of anxiolytics drugs in phobic situations related to the phobia of falling | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  Any change in use of anxiolytics (N05B according to the Anatomical Therapeutic Chemical classification) by participants in phobic situations related to the phobia of falling will be recorded by face-to-face interview.
Self- perceived health | Baseline, 2 months (end of intervention), 5 months (3 month follow-up) and 8 months (6 month follow-up)
  The self-perceived health (SPH) indicator of the Minimum European Health Module is a global measure that encompasses different dimensions of health, i.e. physical, social and emotional function and biomedical signs and symptoms. Self-perceived health appears to be an effective summary of health and has been shown to be a strong predictor of future functional limitations and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine DELPIERRE, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Bretonneau, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided